CLINICAL TRIAL: NCT00927849
Title: Idiopathic Hypertensive Anal Canal: a Place of Internal Sphincterotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: ayman el nakeeb, Mansoura University hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: hypertensive anal canal
Record Dates: First submitted 2009-03-23; First posted 2009-06-25 (Estimated); Results first posted 2009-06-25 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-05

CONDITIONS: Hypertensive Anal Canal
Keywords: anal hypertonia; sphincterotomy; incontinence; manometry
MeSH Terms: interventions — Lateral Internal Sphincterotomy; Nitroglycerin; Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- surgical group lateral sphincterotomy (Active Comparator): underwent closed lateral internal sphincterotomy (LIS) under local anesthesia at 3 o'clock in lithotomy position reaching up to the dentate line.
  Interventions: Procedure: lateral internal sphincterotomy (LIS)
- Glycerin trinitrate group (Active Comparator): all were instructed to apply the Glycerin trinitrate group (GTN) ointment 0.2 % twice a day to the edge and just inside the anal canal for 8 week course.
  Interventions: Drug: Glycerin trinitrate (GTN)
- botulinum toxin injection (Active Comparator): All were injected with botulinum toxin injection (BTX- A) in the left lateral position; anesthesia was not required. A volume of 0.5 ml of dissolved toxin, i.e., 100 u Dysport, is injected in each patient. The injection is given with an insulin syringe fitted with a needle size of 21 gauze and 3.75 lengths. Injection into the IAS, with the patients awake in the left -lateral position in the outpatient clinic in the 3 and 9 o'clock position.
  Interventions: Drug: botulinum toxin injection (BTX A)

INTERVENTIONS:
Procedure: lateral internal sphincterotomy (LIS) — closed lateral internal sphincterotomy was done under local anesthesia at 3 o'clock in lithotomy position reaching up to the dentate line.
  Arms: surgical group lateral sphincterotomy
Drug: Glycerin trinitrate (GTN) — All were instructed to apply the GTN ointment 0.2 % twice a day to the edge and just inside the anal canal for 8 week course.
  Other Names: GTN ointment
  Arms: Glycerin trinitrate group
Drug: botulinum toxin injection (BTX A) — All were injected with botulinum toxin injection (BTX- A) in the left lateral position; anesthesia was not required. A volume of 0.5 ml of dissolved toxin, i.e., 100 u Dysport, is injected in each patient. The injection is given with an insulin syringe fitted with a needle size of 21 gauze and 3.75 lengths. Injection into the IAS, with the patients awake in the left -lateral position in the outpatient clinic in the 3 and 9 o'clock position.
  Other Names: BTX A
  Arms: botulinum toxin injection

SUMMARY:
Idiopathic hypertensive anal canal is a fact and already exists presented by anal pain aggravated by defecation. It can be managed safely by closed lateral sphincterotomy but chemical sphincterotomy had a minor role in its management.

DETAILED DESCRIPTION:
Patient and methods: Sixty three patients complaining of anal pain without any anal pathology and 10 healthy volunteers were examined. All patients underwent clinical evaluation, neurological examination, anorectal manometry, and measurement of pudendal nerve terminal motor latency (PNTML). All patients with hypertensive anal canal were randomized into three groups. Group I (surgical group) underwent closed lateral sphincterotomy LS, group II using nitroglycerine ointment (GTN) and group III received injection of botulinum toxin in internal sphincter. Post procedures data were recorded at follow up period.

ELIGIBILITY:
Inclusion Criteria:

* all patients with hypertensive anal canal

Exclusion Criteria:

* patients who had any pathological anorectal lesions such as anal fissure, piles, rectal prolapse, intussusception, anismus, cancer, patients with normal anal pressure
* patients who previously had anorectal surgery, chemical or surgical sphincterotomy, anal dilatation, IBD, venereal disease, neurological disorder or systemic gastrointestinal disease

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2002-09; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ayman elnakeeb, MD, Principal Investigator — Mansoura University Hospital
Locations (1):
- Ayman Elnakeeb, Al Mansurah, Egypt

REFERENCES:
- [Result] Aysan E, Aren A, Ayar E. A prospective, randomized, controlled trial of primary wound closure after lateral internal sphincterotomy. Am J Surg. 2004 Feb;187(2):291-4. doi: 10.1016/j.amjsurg.2003.11.011. PMID 14769323
- [Result] Brisinda G, Maria G, Bentivoglio AR, Cassetta E, Gui D, Albanese A. A comparison of injections of botulinum toxin and topical nitroglycerin ointment for the treatment of chronic anal fissure. N Engl J Med. 1999 Jul 8;341(2):65-9. doi: 10.1056/NEJM199907083410201. PMID 10395629
- [Result] Orsay C, Rakinic J, Perry WB, Hyman N, Buie D, Cataldo P, Newstead G, Dunn G, Rafferty J, Ellis CN, Shellito P, Gregorcyk S, Ternent C, Kilkenny J 3rd, Tjandra J, Ko C, Whiteford M, Nelson R; Standards Practice Task Force; American Society of Colon and Rectal Surgeons. Practice parameters for the management of anal fissures (revised). Dis Colon Rectum. 2004 Dec;47(12):2003-7. doi: 10.1007/s10350-004-0785-7. No abstract available. PMID 15657647
- [Result] Neill ME, Swash M. Chronic perianal pain: an unsolved problem. J R Soc Med. 1982 Feb;75(2):96-101. doi: 10.1177/014107688207500205. PMID 7069679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: completed , mansoura university hospital
Groups:
- Surgical Group Lateral Sphincterotomy: underwent closed lateral internal sphincterotomy under local anesthesia at 3 o'clock in lithotomy position reaching up to the dentate line.
- Glycein Trinitrate Group: (21) all were instructed to apply the GTN ointment 0.2 % twice a day to the edge and just inside the anal canal for 8 week course.
- Botilinium Toxin Injection: All were injected with BTX- A in the left lateral position; anesthesia was not required. A volume of 0.5 ml of dissolved toxin, i.e., 100 u Dysport, is injected in each patient. The injection is given with an insulin syringe fitted with a needle size of 21 gauze and 3.75 lengths. Injection into the IAS, with the patients awake in the left -lateral position in the outpatient clinic in the 3 and 9 o'clock position.
Period: Overall Study
Arm/Group | Surgical Group Lateral Sphincterotomy | Glycein Trinitrate Group | Botilinium Toxin Injection
Started | 21 | 21 | 21
Completed | 21 | 21 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgical Group Lateral Sphincterotomy | Glycein Trinitrate Group | Botilinium Toxin Injection | Total
Number analyzed (Participants) | 21 | 21 | 21 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 1 | 4.0
  Between 18 and 65 years | 20 | 19 | 20 | 59.0
  >=65 years | 0 | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 41 (5.5) | 40 (7.5) | 40.5 (3.5) | 41 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 16 | 47.0
  Male | 5 | 6 | 5 | 16.0
Region of Enrollment [Number; unit: participants]
  Egypt | 21 | 21 | 21 | 63.0

OUTCOME MEASURES:

1. Primary Outcome: Effect of Closed Lateral Sphincterotomy and Chemical Sphincterotomy on Hypertensive Anal Canal
Description: effect of closed lateral sphincterotomy and chemical sphincterotomy on hypertensive anal canal, anal manometery
Time Frame: one year
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: mmhg

2. Primary Outcome: Relieve of Anal Pain
Description: using a visual analog scale (VAS) with which each patients noted the severity of pain at each evaluated time using a linear between zero (no pain) and 10 ( severe pain)
Time Frame: one year after the procedure
Measure: Mean (Standard Deviation); unit: score in scale
Arm/Group | Surgical Group Lateral Sphincterotomy | Glycein Trinitrate Group | Botilinium Toxin Injection
Number analyzed (Participants) | 21 | 21 | 21
score in scale | 4.16 (2.32) | 4.18 (2.52) | 4.2 (2.42)

ADVERSE EVENTS:
Arm/Group | Surgical Group Lateral Sphincterotomy | Glycein Trinitrate Group | Botilinium Toxin Injection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes